CLINICAL TRIAL: NCT00539981
Title: Evaluation of the Immunogenicity, Safety, Reactogenicity, Efficacy, Effectiveness and Lot Consistency of FluBlok® Trivalent Recombinant Baculovirus-Expressed Hemagglutinin Influenza Vaccine in Healthy Adults Aged 18 to 49 Years
Brief Title: Immunogenicity, Safety, Reactogenicity, Efficacy, Effectiveness and Lot Consistency of FluBlok
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Protein Sciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PSC04
Record Dates: First submitted 2007-10-03; First posted 2007-10-05 (Estimated); Results first posted 2021-02-15 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — FluBlok

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FluBlok (Lots A, B, C) (Experimental): Participants received a single 0.5 milliliters (mL) dose of FluBlok vaccine from any of the Lots A, B, or C, intramuscularly on Day 0 (Visit 1). Participants were followed up to 6 months after vaccination.
  Interventions: Biological: FluBlok®
- Placebo (Placebo Comparator): Participants received a single dose of placebo matched to FluBlok, intramuscularly on Day 0 (Visit 1). Participants were followed up to 6 months after vaccination.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: FluBlok® — Dose: 0.5 mL, single dose; Route of administration: intramuscular. Recombinant Trivalent Hemagglutinin Influenza Vaccine containing 45 microgram (mcg) of each hemagglutinin derived from A/Solomon Islands/3/2006 (H1N1), A/Wisconsin/67/2005 (H3N2), and B/Malaysia/2506/2004
  Other Names: rHA Trivalent Recombinant Hemagglutinin Influenza Vaccine
  Arms: FluBlok (Lots A, B, C)
Biological: Placebo — Dose: 0.5 mL normal saline for injection, single dose; Route of administration: intramuscular
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate a single dose of FluBlok in terms of safety, efficacy and effectiveness in prevention of influenza and influenza-like illness and assess clinical lot-to-lot consistency in manufacturing by evaluating and comparing the immunogenicity of three different lots of FluBlok in a subset of participants.

DETAILED DESCRIPTION:
All currently licensed influenza vaccines in the United States were produced in embryonated hen's eggs. There were several well-recognized disadvantages to the use of eggs as the substrate for influenza vaccine. Eggs required specialized manufacturing facilities and could be difficult to scale up rapidly in response to an emerging need such as a pandemic. It was usually necessary to adapt candidate vaccine viruses for high-yield growth in eggs, a process that could be time consuming, was not always successful, and could select receptor variants that might have suboptimal immunogenicity. In addition, agricultural diseases that affected chicken flocks, and that might be an important issue in a pandemic due to an avian influenza virus strain, could easily disrupt the supply of eggs for vaccine manufacturing. Therefore, development of alternative substrates for influenza vaccine production had been identified as a high-priority objective.

One potential alternative method for production of influenza vaccine was expression of the influenza virus hemagglutinin (HA) using recombinant deoxyribonucleic acid (DNA) techniques. This alternative avoided dependence on eggs and was very efficient because of the high levels of protein expression under the control of the baculovirus polyhedrin promoter.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18-49 years.
* Provided informed consent prior to any study procedures.
* Able to comply with all study procedures.
* Available for follow-up for the duration of the influenza season.
* Women of child-bearing potential must have had a negative urine pregnancy test at the time of randomization and must be willing to use an adequate form of contraception (includes abstinence, condom with spermicide, licensed hormonal contraceptive, intrauterine device [IUD], monogamous relationship with a vasectomized partner) during the course of the study.

Exclusion Criteria:

* Long-term use of oral steroids, parenteral steroids, or high-dose inhaled steroids (greater than [>] 800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (Nasal and topical steroids were allowed).
* Presence of high-risk conditions or other characteristics were considered to be indication for influenza vaccination, as defined by the Advisory Committee on Immunization Practices.
* Acute febrile illness (defined as having a temperature greater than or equal to [>=]100 degrees Fahrenheit) or upper respiratory tract illness within 72 hours of vaccination. Participants with acute febrile illness were rescheduled after fever resolved.
* Use of experimental vaccines or any influenza vaccine other than FluBlOk after May 31st 2007 for the 2008 Southern Hemisphere or 2007 to 2008 Northern hemisphere epidemic seasons.
* Immunosuppression as a result of an underlying illness or treatment, or used anticancer chemotherapy or radiation therapy within the preceding 36 months.
* Any malignancy diagnosed or treated actively during the past five (5) years, with two (2) exceptions. Participant with any history of lymphoproliferative disorder were excluded. However, participants with a history of localized non-melanotic skin cancer were eligible.
* Receipt of any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study.
* Receipt of an experimental agent (vaccine, drug, biologic, device, blood product or medication) within 1 month prior to enrollment in this study, or expected to receive an experimental agent during study period.
* Receipt of parenteral immunoglobulin or other blood product within the three months prior to study vaccination.
* Major psychiatric diagnosis including schizophrenia, bipolar disease or other major depression, or any diagnosis of dementia or associated concomitant medications (e.g., Aricept) used for treating dementia.
* Known active human immunodeficiency virus, hepatitis B, or hepatitis C infection.
* History of alcohol or drug abuse in the last 5 years.
* Not available for three or more consecutive weeks during flu surveillance period.
* Any acute or chronic condition that, in the opinion of the investigator, would render vaccination unsafe or interfere with the evaluation of responses or render the participant unable to meet the requirements of the protocol.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4648 (Actual)
Dates: Start 2007-09-15 (Actual); Primary Completion 2008-05-28 (Actual); Study Completion 2008-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J Treanor, MD, Principal Investigator — University of Rochester
Locations (24):
- United States (24):
  - Impact Clinical Trials, Beverly Hills, California
  - Benchmark Research - Sacramento, Sacramento, California
  - Benchmark Research - San Francisco, San Francisco, California
  - University Clinical Research, Inc, Pembroke Pines, Florida
  - Vince and Associates, Overland Park, Kansas
  - Kentucky pediatric /Adult Research, Bardstown, Kentucky
  - Benchmarch Research - New Orleans, Metairie, Louisiana
  - University of Maryland - Baltimore, Baltimore, Maryland
  - Saint Louis University, St Louis, Missouri
  - Meridian Clinical Research, Omaha, Nebraska
  - Regional Clinical Research, Inc., Endwell, New York
  - Rochester Medical Center, Rochester, New York
  - Carolina Medical Trials, Winston-Salem, North Carolina
  - Sterling Research, Cincinnati, Ohio
  - Primary Physicians Research - Pediatric Alliance St. Clair, Pittsburgh, Pennsylvania
  - Primary Physicians Research, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Benchmarch Research - Austin, Austin, Texas
  - Benchmark Research - Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Benchmark Research - San Angelo, San Angelo, Texas
  - Jean Brown Research, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Marshfield Clinic, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Background] Treanor JJ, El Sahly H, King J, Graham I, Izikson R, Kohberger R, Patriarca P, Cox M. Protective efficacy of a trivalent recombinant hemagglutinin protein vaccine (FluBlok(R)) against influenza in healthy adults: a randomized, placebo-controlled trial. Vaccine. 2011 Oct 13;29(44):7733-9. doi: 10.1016/j.vaccine.2011.07.128. Epub 2011 Aug 9. PMID 21835220
- [Derived] Rajendran M, Nachbagauer R, Ermler ME, Bunduc P, Amanat F, Izikson R, Cox M, Palese P, Eichelberger M, Krammer F. Analysis of Anti-Influenza Virus Neuraminidase Antibodies in Children, Adults, and the Elderly by ELISA and Enzyme Inhibition: Evidence for Original Antigenic Sin. mBio. 2017 Mar 21;8(2):e02281-16. doi: 10.1128/mBio.02281-16. PMID 28325769
- [Derived] Nachbagauer R, Choi A, Izikson R, Cox MM, Palese P, Krammer F. Age Dependence and Isotype Specificity of Influenza Virus Hemagglutinin Stalk-Reactive Antibodies in Humans. mBio. 2016 Jan 19;7(1):e01996-15. doi: 10.1128/mBio.01996-15. PMID 26787832
- See also: Related Info — http://proteinsciences.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 24 active centers in the United States from 15-September-2007 to 28-May-2008.
Pre-assignment Details: A total of 4648 participants were randomized in the study. Participants were randomized in 1:1 ratio to receive FluBlok or Placebo. The FluBlok assignment was further stratified into three lots, A, B and C to assess lot consistency.
Period: Overall Study
Arm/Group | FluBlok (Lots A, B, C) | Placebo
Started | 2344 | 2304
Completed | 2049 | 2022
Not Completed | 295 | 282
Not completed — Adverse events (AE) | 3 | 3
Not completed — Lost to Follow-up | 260 | 251
Not completed — Withdrew consent | 22 | 14
Not completed — Death | 1 | 1
Not completed — Other reason-unspecified | 9 | 13

BASELINE CHARACTERISTICS:
Population: Analysis performed on safety population that included participants who received study vaccine, according to the treatment (FluBlok or Placebo) actually received.
Groups:
- FluBlok (Lots A, B, C): Participants received a single 0.5 mL dose of FluBlok vaccine from any of the Lots A, B, or C, intramuscularly on Day 0 (Visit 1). Participants were followed up to 6 months after vaccination.
- Total: Total of all reporting groups
Arm/Group | FluBlok (Lots A, B, C) | Placebo | Total
Number analyzed (Participants) | 2344 | 2304 | 4648
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2344 | 2304 | 4648
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1391 | 1349 | 2740
  Male | 953 | 955 | 1908
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White/Caucasian | 1570 | 1530 | 3100
  Race/Ethnicity: Black/African-American | 430 | 447 | 877
  Race/Ethnicity: Latino/Hispanic | 250 | 239 | 489
  Race/Ethnicity: Asian | 62 | 52 | 114
  Race/Ethnicity: American Indian/Alaska Native | 7 | 9 | 16
  Race/Ethnicity: Native Hawaiian/Pacific Islander | 6 | 8 | 14
  Race/Ethnicity: Other-unspecified | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Solicited Injection Site (Local) Reactions
Description: Solicited reaction (reactogenicity event) was an adverse event (AE) that was pre-listed in electronic case report form(eCRF), considered to be related to vaccination and recorded by participant by means of memory aid. Injection sites reaction included pain,bruising,redness,swelling. Pain and bruising:Grade0: didn't have it at all; Grade1: noticed it, but it didn't interfere with usual activities at all; Grade2: had it, and it was bad enough to prevent a significant part of usual activities; Grade3: had it, and it prevented most or all of normal activities, or had to see a doctor for prescription medicine, Redness and swelling: participants measured largest diameter of any injection site reaction and grade them from 0 to 3, where Grade0: measured less than(<)10 milliliters(mm); Grade1: larger than or equal to(>=) 10mm and <20mm; Grade 2: >=20mm and <50mm; Grade3: >=50mm. Participants with multiple symptoms in same category were counted once per category using symptom with maximum grade
Time Frame: Within 7 days post vaccination
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | FluBlok (Lots A, B, C) | Placebo
Number analyzed (Participants) | 2344 | 2304
Participants
  Injection site pain- Grade 0 | 1421 | 2050
  Injection site pain- Grade 1 | 797 | 177
  Injection site pain- Grade 2 | 52 | 3
  Injection site pain- Grade 3 | 2 | 1
  Injection site bruising- Grade 0 | 2197 | 2172
  Injection site bruising- Grade 1 | 68 | 57
  Injection site bruising- Grade 2 | 6 | 1
  Injection site bruising- Grade 3 | 1 | 1
  Injection site redness- Grade 0 | 2181 | 2184
  Injection site redness- Grade 1 | 72 | 40
  Injection site redness- Grade 2 | 15 | 6
  Injection site redness- Grade 3 | 4 | 1
  Injection site swelling- Grade 0 | 2195 | 2189
  Injection site swelling- Grade 1 | 55 | 34
  Injection site swelling- Grade 2 | 16 | 6
  Injection site swelling- Grade 3 | 6 | 2

2. Primary Outcome: Number of Participants Reporting Solicited Systemic Reactions
Description: Solicited reaction (reactogenicity event) was an AE that was pre-listed in eCRF, considered to be related to vaccination recorded by the participant by means of a memory aid between the day of vaccination (Day 0) and Day 7 post vaccination. Systemic events included fever, fatigue, shivering, joint pain, muscle pain, headache, and nausea. Fever: >=100.4 degree Fahrenheit (ºF) to <101.1ºF; >=101.2ºF to <102.2ºF; >=102.2ºF; Fatigue, shivering, joint pain, muscle pain, headache and nausea: Grade 0: didn't have it at all; Grade 1: noticed it, but it didn't interfere with usual activities at all; Grade 2: had it, and it was bad enough to prevent a significant part of usual activities; and Grade 3: had it, and it prevented most or all of normal activities, or had to see a doctor for prescription medicine. Participants with multiple symptoms in the same category were counted once per category using the symptom with the maximum grade.
Time Frame: Within 7 days post vaccination
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | FluBlok (Lots A, B, C) | Placebo
Number analyzed (Participants) | 2344 | 2304
Participants
  Fever (>=100.4ºF) | 2238 | 2188
  Fever (>=100.4 to <101.1ºF) | 8 | 5
  Fever (>=101.2 to <102.2ºF) | 5 | 6
  Fever (>=102.2ºF) | 4 | 1
  Fatigue- Grade 0 | 1932 | 1898
  Fatigue- Grade 1 | 250 | 256
  Fatigue- Grade 2 | 78 | 66
  Fatigue- Grade 3 | 12 | 11
  Shivering- Grade 0 | 2202 | 2160
  Shivering- Grade 1 | 52 | 54
  Shivering- Grade 2 | 12 | 13
  Shivering- Grade 3 | 6 | 4
  Joint pain- Grade 0 | 2183 | 2148
  Joint pain- Grade 1 | 69 | 67
  Joint pain- Grade 2 | 14 | 12
  Joint pain- Grade 3 | 6 | 4
  Muscle pain- Grade 0 | 2033 | 2077
  Muscle pain- Grade 1 | 197 | 124
  Muscle pain- Grade 2 | 36 | 22
  Muscle pain- Grade 3 | 6 | 8
  Headache- Grade 0 | 1923 | 1877
  Headache- Grade 1 | 264 | 273
  Headache- Grade 2 | 70 | 68
  Headache- Grade 3 | 15 | 13
  Nausea- Grade 0 | 2143 | 2122
  Nausea- Grade 1 | 94 | 74
  Nausea- Grade 2 | 29 | 25
  Nausea- Grade 3 | 6 | 10

3. Primary Outcome: Number of Participants Reporting Unsolicited Adverse Events
Description: An AE was defined as any unfavorable and unintended sign (e.g., a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a study vaccine, whether or not considered to be related to the study vaccine. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted (i.e., solicited) in the eCRF in terms of symptom and/or onset post-vaccination, ascertained during follow-up visit or telephone contact up to (and including) the Day 28 contact, whether reported spontaneously by the participant or in response to general questions about current or interim health status.
Time Frame: From Day 0 (post-vaccination) through Day 28 post vaccination
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | FluBlok (Lots A, B, C) | Placebo
Number analyzed (Participants) | 2344 | 2304
Participants | 61 | 67

4. Primary Outcome: Lot Consistency: Geometric Mean Titers (GMTs) of Influenza Vaccine Antibodies Following FluBlok Vaccination
Description: GMTs of anti-influenza antibodies were measured using a single radial immunodiffusion (SRID) assay for 3 strains: A/Solomon Islands [H1N1], A/Wisconsin [H3N2], and B/Malaysia. Titers were expressed in terms of 1/dilution.
Time Frame: Day 28 post vaccination
Population: Analysis was done on evaluable population that included all participants who had met the study entry criteria and had titers taken at Baseline (Day 0) and after vaccination (Day 28). Data for this outcome measure was planned to be collected and analyzed for each FluBlok lot separately and not planned to be collected for placebo, as pre-specified in protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer (1/dilution)
Groups:
- FluBlok: Lot A: Participants received a single 0.5 mL dose of FluBlok vaccine from Lot A, intramuscularly on Day 0 (Visit 1). Participants were followed up to 6 months after vaccination.
- FluBlok: Lot B: Participants received a single 0.5 mL dose of FluBlok vaccine from Lot B, intramuscularly on Day 0 (Visit 1). Participants were followed up to 6 months after vaccination.
- FluBlok: Lot C: Participants received a single 0.5 mL dose of FluBlok vaccine from Lot C, intramuscularly on Day 0 (Visit 1). Participants were followed up to 6 months after vaccination.
Arm/Group | FluBlok: Lot A | FluBlok: Lot B | FluBlok: Lot C
Number analyzed (Participants) | 150 | 151 | 147
Titer (1/dilution)
  A/Solomon Islands (H1N1) | 346.15 [291.96 to 410.41] | 322.95 [274.80 to 379.55] | 381.00 [321.79 to 451.10]
  A/Wisconsin (H3N2) | 390.34 [324.83 to 469.06] | 192.25 [159.59 to 231.59] | 240.01 [200.14 to 287.82]
  B/Malaysia | 182.10 [151.95 to 218.24] | 205.95 [174.16 to 243.55] | 215.34 [179.31 to 258.62]
Statistical Analysis 1: Comparison: FluBlok: Lot A vs FluBlok: Lot B; A/Solomon Islands (H1N1): FluBlok: Lot A versus FluBlok: Lot B; Test type: Equivalence — Equivalence between 2 lots for each strain was concluded if the 2-sided 95% CI for the ratio of post-vaccination GMTs for Lot A vs. B falls within 0.67 to 1.5; p = 0.009, ANOVA — Threshold for significance of p value was 0.05; GMT ratio = 1.07, 95% CI 2-sided [0.85 to 1.36]
Statistical Analysis 2: Comparison: FluBlok: Lot A vs FluBlok: Lot C; A/Solomon Islands (H1N1): FluBlok: Lot A versus FluBlok: Lot C; Test type: Equivalence — Equivalence between 2 lots for each strain was concluded if the 2-sided 95% CI for the ratio of post-vaccination GMTs for Lot A vs. C falls within 0.67 to 1.5; p = 0.009, ANOVA — Threshold for significance of p value was 0.05; GMT ratio = 0.91, 0.91% CI 2-sided [0.71 to 1.15]
Statistical Analysis 3: Comparison: FluBlok: Lot B vs FluBlok: Lot C; A/Solomon Islands (H1N1): FluBlok: Lot B versus FluBlok: Lot C; Test type: Equivalence — Equivalence between 2 lots for each strain was concluded if the 2-sided 95% CI for the ratio of post-vaccination GMTs for Lot B vs. C falls within 0.67 to 1.5; p = 0.009, ANOVA; Threshold for significance of p value was 0.05; GMT ratio = 0.85, 95% CI 2-sided [0.67 to 1.07]
Statistical Analysis 4: Comparison: FluBlok: Lot A vs FluBlok: Lot B; A/Wisconsin (H3N2): FluBlok: Lot A versus FluBlok: Lot B; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; p = 0.065, ANOVA — Threshold of significance for p value was 0.05; GMT ratio = 2.03, 95% CI 2-sided [1.56 to 2.64]
Statistical Analysis 5: Comparison: FluBlok: Lot A vs FluBlok: Lot C; A/Wisconsin (H3N2): FluBlok: Lot A versus FluBlok: Lot C; Test type: Equivalence — [test comment as in outcome 4, analysis 2]; p = 0.065, ANOVA; Threshold of significance for p value was 0.05; GMT ratio = 1.63, 95% CI 2-sided [1.26 to 2.11]
Statistical Analysis 6: Comparison: FluBlok: Lot B vs FluBlok: Lot C; A/Wisconsin (H3N2): FluBlok: Lot B versus FluBlok: Lot C; Test type: Equivalence — [test comment as in outcome 4, analysis 3]; p = 0.065, ANOVA; Threshold of significance for p value was 0.05; GMT ratio = 0.80, 95% CI 2-sided [0.62 to 1.04]
Statistical Analysis 7: Comparison: FluBlok: Lot A vs FluBlok: Lot B; B/Malaysia: FluBlok: Lot A versus FluBlok: Lot B; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; p = 0.011, ANOVA; Threshold of significance for p value was 0.05; GMT ratio = 0.88, 95% CI 2-sided [0.69 to 1.13]
Statistical Analysis 8: Comparison: FluBlok: Lot A vs FluBlok: Lot C; B/Malaysia: FluBlok: Lot A versus FluBlok: Lot C; Test type: Equivalence — [test comment as in outcome 4, analysis 2]; p = 0.011, ANOVA; Threshold of significance for p value was 0.05; GMT ratio = 0.85, 95% CI 2-sided [0.65 to 1.09]
Statistical Analysis 9: Comparison: FluBlok: Lot B vs FluBlok: Lot C; B/Malaysia: FluBlok: Lot B versus FluBlok: Lot C; Test type: Equivalence — [test comment as in outcome 4, analysis 3]; p = 0.011, ANOVA; Threshold of significance for p value was 0.05; GMT ratio = 0.96, 95% CI 2-sided [0.75 to 1.23]

5. Primary Outcome: Percentage of Participants With Positive Cell Culture/Culture-Confirmed Influenza Like Illness as Defined by Centers for Disease Control and Prevention (CDC-ILI)
Description: CDC-defined ILI was defined as fever (body temperature >=100ºF oral accompanied by cough and/or sore throat, on the same day or on consecutive days) due to strains represented in the vaccine.
Time Frame: 14 days post vaccination through and up to 6 months
Population: Analysis was performed on safety population.
Measure: Number; unit: percentage of participants
Arm/Group | FluBlok (Lots A, B, C) | Placebo
Number analyzed (Participants) | 2344 | 2304
percentage of participants | 0.04 | 0.2
Statistical Analysis 1: Comparison: FluBlok (Lots A, B, C) vs Placebo; FluBlok versus Placebo; Test type: Superiority — Relative protective efficacy is equivalent to absolute efficacy which is defined as the reduction in the influenza rate for Flublok relative to placebo; Relative protective efficacy = 75.4, 95% CI 2-sided [-148.0 to 99.5]

6. Secondary Outcome: Percentage of Participants With Seroprotection to Influenza Vaccine Antigens After Vaccination With FluBlok
Description: Anti-influenza antibodies were measured using an HAI assay for 3 strains: A/Solomon Islands [H1N1], A/Wisconsin [H3N2] and B/Malaysia. Seroprotection was defined as a post-vaccination HAI antibody titer of >=1:40.
Time Frame: 28 days post vaccination
Population: Analysis was performed on evaluable population. Data for this outcome measure was not planned to be collected and analyzed for placebo group, as pre-specified in protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FluBlok (Lots A, B, C)
Number analyzed (Participants) | 448
percentage of participants
  A/Solomon Islands (H1N1) | 99 [97.1 to 99.5]
  A/Wisconsin (H3N2) | 97 [94.8 to 98.3]
  B/Malaysia | 96 [94.0 to 97.8]

7. Secondary Outcome: Percentage of Participants With Seroconversion to Influenza Vaccine Antigens After Vaccination With FluBlok
Description: Anti-influenza antibodies were measured using an HAI assay for 3 strains: A/Solomon Islands [H1N1], A/Wisconsin [H3N2] and B/Malaysia. Seroconversion was defined as a post-vaccination titer of >=1:40 in participants with undetectable baseline antibody (HI titer = <1:10) or a >=4-fold rise in antibody in participants with a baseline titer of >=1:10, with the achievement of post-vaccination titer of at least 1:40.
Time Frame: 28 days post vaccination
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FluBlok (Lots A, B, C)
Number analyzed (Participants) | 448
percentage of participants
  A/Solomon Islands (H1N1) | 78 [73.5 to 81.5]
  A/Wisconsin (H3N2) | 81 [77.1 to 84.6]
  B/Malaysia | 52 [47.0 to 56.5]

ADVERSE EVENTS:
Time Frame: Unsolicited non-serious AEs: Day 0 to Day 28 post vaccination, Solicited reactions: within 7 days post vaccination, SAE: through the end of influenza season (up to 6 months)
Description: Solicited reaction was AE that was prelisted (i.e., solicited) in the eCRF and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted (i.e., solicited) in the eCRF in terms of symptom and/or onset post-vaccination. Analysis was performed on Safety population.
Arm/Group | FluBlok (Lots A, B, C) | Placebo
All-Cause Mortality (participants affected / at risk) | 1/2344 | 1/2304
Serious Adverse Events (participants affected / at risk) | 30/2344 | 34/2304
Other Adverse Events (participants affected / at risk) | 152/2344 | 120/2304
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FluBlok (Lots A, B, C) (N=2344) | Placebo (N=2304)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Rathke's cleft cyst (Congenital, familial and genetic disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Accidental death (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 2
Cellulitis (Infections and infestations) | 0 | 1
Hepatitis viral (Infections and infestations) | 1 | 0
Infected insect bite (Infections and infestations) | 0 | 1
Infectious mononucleosis (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 0 | 2
Perianal abscess (Infections and infestations) | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Postoperative infection (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Staphylococcal abscess (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0
Open fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 1
Aseptic necrosis bone (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Headache (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Pregnancy induced hypertension (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Adjustment disorder (Psychiatric disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 3
Suicidal ideation (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 2 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Adnexa uteri mass (Reproductive system and breast disorders) | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 1
Dyspareunia (Reproductive system and breast disorders) | 0 | 1
Endometrial disorder (Reproductive system and breast disorders) | 1 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Prolapsed bladder (Reproductive system and breast disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FluBlok (Lots A, B, C) (N=2344) | Placebo (N=2304)
Headache (Nervous system disorders) | 35 | 42
Cough (Respiratory, thoracic and mediastinal disorders) | 48 | 37
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 37 | 31
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 42 | 49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.